CLINICAL TRIAL: NCT03758833
Title: Single or Double Elective Embryos Transfer Associated to Preimplantation Genetic Test in in Vitro Fertilization Cycles
Brief Title: eSET or eDET Associated to PGT in IVF
Acronym: SetDetPgt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Pedro Augusto Araújo Monteleone, Clinical Head of the Reproductive Medicine Center Governador Mario Covas, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SET-NGS
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: in Vitro Fertilization; Single Embryo Transfer; Preimplantation Genetic Diagnosis; Pregnancy
Keywords: in vitro fertilization; single embryo transfer; preimplantation genetic diagnosis; clinical pregnancy
MeSH Terms: interventions — Single Embryo Transfer; DEET

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SET (Active Comparator): patients receiving the elective single embryo transfer
  Interventions: Procedure: Single embryo transfer
- SET+NGS (Experimental): patients receiving the elective single embryo transfer evaluated genetically by NGS
  Interventions: Diagnostic Test: preimplantation genetic test of embryo by new generation sequencing (NGS); Procedure: Single embryo transfer
- DET (Active Comparator): patients receiving the elective double embryo transfer
  Interventions: Procedure: Double embryo tranfer
- DET+NGS (Experimental): patients receiving the elective double embryo transfer evaluated genetically by NGS
  Interventions: Diagnostic Test: preimplantation genetic test of embryo by new generation sequencing (NGS); Procedure: Double embryo tranfer

INTERVENTIONS:
Diagnostic Test: preimplantation genetic test of embryo by new generation sequencing (NGS) — This is a genetic test to evaluate 24 chromosomes by the new generation sequencing platform. For that is necessary a embryo biopsy in the blastocyst stage and evaluation of a greater number of cells extracted from the trophectoderm
  Arms: DET+NGS; SET+NGS
Procedure: Single embryo transfer — Transfer of single embryo
  Other Names: SET
  Arms: SET; SET+NGS
Procedure: Double embryo tranfer — Transfer of two embryos
  Other Names: DET
  Arms: DET; DET+NGS

SUMMARY:
In vitro fertilization (IVF) techniques have been improving performance recently and, nowadays, provide a live birth rate of around 25%. The success of IVF techniques is dependent upon maximum efficiency at each stage of treatment, and, at the same time, high success rates with a low risk of complications. Multiple pregnancies are one of the most important adverse event of IVF techniques. In this sense, the use of elective single embryo transfer (SET) has become an option for patients with good prognosis compared to the transfer of multiple embryos, and it is recommended in order to reduce the risk of multiple pregnancies and their consequences. On the other hand, it is known that embryonic quality is a crucial step for the success of IVF techniques and the efficiency of this process is linked to the decrease in the number of embryos to be transferred. Usually, embryo selection is based on morphological and developmental criteria. However, recently, it has been demonstrated that the blastocyst biopsy associated with the chromosomal / genetic screening may be a predictor of the chances of implantation. The investigators group demonstrated the feasibility of performing SET sequentially, promoting satisfactory gestation rates and safety for the mother and baby regarding multiple gestation for patients with good prognosis. Based on these principles, the investigators raised the hypothesis that SET associated with preimplantation genetic diagnosis (PGD) by next-generation sequencing (NGS) for patients with good prognosis can improve the success rates of IVF cycles and, at the same time, avoid multiple pregnancies, as well as maternal-fetal and neonatal risks resulting from this condition. To test this hypothesis, the aim of this study is to compare the results of IVF treatments in patients receiving SET (SET group), SET associated with genetic evaluation by NGS (group NGS + SET), elective transference of two embryos (DET group) and DET associated with genetic evaluation by NGS (NGS + DET). In case of non-pregnancy on the first transfer, there will be subsequent transfers until the remaining embryos are exhausted or the patient reaches the gestation. The primary endpoint will be the cumulative pregnancy rate per treatment cycle and this approach will allow to confirm or not the hypothesis that genetic analysis is effective in improving the embryo selection process and associated with SET will increase clinical gestation rates and decrease rates of multiple gestations and miscarriages.

DETAILED DESCRIPTION:
Infertility is an important public health problem, affecting between 8 and 12% of reproductive-age couples, and leading to a high prevalence of childless couples (Bergstrom, 1992; Ombelet and Campo, 2007). The demand for infertility treatment is increasing due to sociocultural factors such as delayed pregnancy, higher incidence of sexually transmitted diseases, obesity rates, and greater acceptance to the available treatments. Recent estimates have shown that more than 1.8 million assisted reproduction treatments (ART) were performed in 2010 and more than 6 million children born were conceived using ART (Dyer et al., 2016).

In vitro fertilization (IVF) techniques have improved performance and currently provide a live embryo transfer rate that is around 25%. However, the success of IVF techniques depends on maximum efficiency in each treatment step, from controlled ovarian stimulation to obtaining adequate numbers of good quality mature eggs, optimal embryo culture conditions, availability of embryos of good quality for transfer and an adequate endometrium for implantation. Changes in clinical and laboratory practices such as the transfer of embryos in the blastocyst stage, improvement of cryopreservation techniques, transfer of thawed embryos after endometrial preparation and single embryo transfer (SET), have been increasingly indicated for patients with good prognosis. At the same time, the use of SET and freezing of all embryos for later transfer of thawed embryos are the major paradigms of ART in recent years (Chambers et al., 2016).

Despite a variation among countries influenced by coverage of health plans, legislation, guides to medical societies, population and culture, in Europe, on average 20% of transfers are single, with up to 69% of cycles in Sweden. In the United States, elective SET is still low, around 10% among women up to 35 years of age (Maheshwari et al., 2011; Practice Committee of the Society for Assisted Reproductive and Practice Committee of the American Society for Reproductive Medicine, 2012). Despite recommendations and increased SET practice, multiple gestation rates in IVF techniques are still high in the overall mean, around 20-25%, as a result of resistance of using SET and maintaining the transfer of multiple embryos with the purpose of obtaining higher gestation rates (Naasan et al., 2012, Kupka et al., 2014, Ishihara et al., 2015). This resistance is due to the idea that transferring more than one embryo may increase the chance of gestation. However, this practice does not take in consideration the increase of maternal and perinatal complications due to multiple pregnancies (Min et al., 2010; Practice Committee of American Society for Reproductive, 2012). In addition, studies have shown that cumulative live birth rates after the transfer of two SET cycles are comparable with a single transfer of two embryos (Pandian et al., 2009; Chambers and Ledger, 2014).

Historically, it is known that among the total number of retrieved oocytes, only a limited amount of them carry the potential to generate full-term gestation. Thus, embryo selection is a crucial step for the success of IVF techniques and the efficiency of this process is related to the decrease in the number of embryos to be transferred, since once it is possible to select embryos with greater implantation potential, the transfer of fewer embryos becomes more feasible and effective. In the routine, the embryonic selection is based on morphological criteria and characteristics of embryo development in order to infer its implantation potential (Ebner et al., 2003).

After controlled ovarian stimulation, approximately 50% of the embryos present chromosomal alterations (Munne et al., 1995). Then, the embryonic genetic evaluation is becoming increasingly used for the selection of euploid embryos for transfer. Blastocyst biopsy associated with chromosomal screening has been shown to be highly predictive of blastocyst developmental potential (Scott et al., 2012), increasing the chances of implantation by selection of euploid blastocysts for transfer in fresh (Scott et al., 2013) and frozen-thawed cycles (Schoolcraft and Katz-Jaffe, 2013).

In addition, preimplantation genetic screening (PGS) is indication for advanced maternal age (Schoolcraft et al., 2009), repeated implantation failure (Blockeel et al., 2008; Rubio et al. 2013), repeat miscarriage (Shahine and Lathi, 2014) and severe male factor (Harper and Sengupta, 2012). More recently, the use of PGS in cases of good prognosis for embryo selection in SET cycles has been proposed for both young and good prognosis patients (Yang et al., 2012), as well as for those in advanced age (Schoolcraft and Katz -Jaffe, 2013), with an important increase in the rate of embryo transfer associated with a reduction in the rates of multiple gestation (Ubaldi et al., 2015).

PGD was initially performed by in fluorescent in situ hybridization (FISH) technology from embryo biopsy on the third day of the development and analysis of one or two blastomeres by evaluating a limited number of chromosomes. The evolution of this technology led to the complete analysis of the 24 chromosomes by the comparative genome hybridization (CGH) platform associated with embryo biopsy in the blastocyst stage and evaluation of a greater number of cells extracted from the trophectoderm. This approach is associated with higher rates of clinical gestation, improved embryo selection in SET cycles and decreasing multiple gestations in patients with good prognosis (Dahdouh et al., 2015). More recently, the next-generation sequencing (NGS) platform has been used and validated for embryonic genetic analysis in IVF, which is used for whole genome amplification (WGA), with the advantage of being a technology with potential to improve the embryonic chromosomal diagnosis in terms of robustness, automation and ability to detect aneuploidies (Fiorentino et al., 2014; Wells et al., 2014).

A recent study developed by the investigators group suggests that patients with good prognosis who perform SET in a fresh cycle and did not become pregnant, do not benefit from receiving a second transfer of two embryos, since the gestation rates are similar to those of patients who received one embryo in the second transfer, with the disadvantage of having a high incidence of multiple pregnancies. These results obtained in a retrospective study already indicate the advantages of performing SET in a sequential manner, promoting satisfactory gestation rates and safety for the mother and baby with regard to multiple gestation for patients with good prognosis (Monteleone et al. , 2016).

Based on these principles, the investigators consider that elective single embryo transfer (SET) associated with preimplantation genetic diagnosis by NGS (NGS + SET) for patients with good prognosis can result in higher success rates of IVF cycles and at the same time decreases multiple pregnancies, as well as maternal-fetal and neonatal risks inherited from this condition. This protocols is suppose to result in high rates of clinical gestation with less occurrence of abortions and greater overall success of the treatment. In order to prove this hypothesis, the investigators propose a study that compares the outcomes of IVF treatments in patients receiving the elective transfer of single embryo genetically evaluated by NGS (NGS + SET) and elective transference of two embryos genetically evaluated by NGS (NGS + DET). As a control, this study will include embryo transfer groups without preimplantation genetic diagnosis by NGS, that is, those that are selected for transfer only from morphological criteria as routine, being associated also the elective transference of one (SET) or two embryos (DET). In case of non-pregnancy in the first cycle of IVF, there will be subsequent transfers of one or two embryos respectively for each group until the remaining embryos are exhausted or until the patient reaches the gestation. The primary outcome will be the cumulative pregnancy rate per treatment cycle. This approach will allow to confirm or not the hypothesis that genetic analysis is effective in improving the embryo selection process and associated with SET will increase the rates of clinical gestation and decrease the rates of multiple gestations and miscarriages.

ELIGIBILITY:
Inclusion Criteria:

* Couples performing in vitro fertilization cycles using intracytoplasmic sperm injection

  * Performing the first treatment cycle;
  * Body Mass Index (BMI) of 18 to 30 kg / m2;
  * Presence of both ovaries without evidence of significant abnormalities;
  * Absence of any significant pathology of the endometrial cavity, such as polyps, fibroids larger than 4cm and hidrosalpinge;
  * Normal ovarian reserve, determined by antral follicle count> 8 and FSH <12 mIU / mL;
  * Use of fresh ejaculate or cryopreserved partner seminal sample

Exclusion Criteria:

* Women presenting endometriosis degrees III and IV;

  * Sperm used for fertilization from partner with severe oligozoospermia (<5 million sperm / ml);
  * Women with associated systemic diseases or infectious diseases;
  * Do not have at least two good quality blastocysts on the fifth day of development.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
cumulative pregnancy rate | 6 months
  percentage of patients who become pregnant after transfer of embryos

SECONDARY OUTCOMES:
cycle cancellation rate | 1 month
  percentage of cycles cancelled due to all embryos genetic alterated
multiple pregnancy rate | 6 months
  percentage of patients who become pregnant of twins
live birth rates | one year
  percentage of patients who had live birth
transfers needed to achieve gestation | 6 months
  number of embryos transfers needed to achieve gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade de São Paulo (FMUSP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No